CLINICAL TRIAL: NCT06513442
Title: The Added Value of Bone Microstructure Assessment in the Management of Osteoporotic Bone
Acronym: ADVANTAGE BONE
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1.1
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trabecular bone score software — To assess the clinical utility of trabecular bone score (TBS) on fracture risk prediction including the new version (TBS V4) and future TBS versions at the spine and hip.

SUMMARY:
1. To assess the clinical utility of trabecular bone score (TBS) on fracture risk prediction including the new version (TBS V4) and future TBS versions at the spine and hip.
2. To assess the clinical utility of TBS software as a potential treatment outcome: sensitivity to change over time and following osteoporosis therapy.
3. To compare TBS to other imaging modalities of bone structure such as quantitative computed tomography (QCT) in fracture risk prediction and response to osteoporosis therapy.

ELIGIBILITY:
Inclusion Criteria: Has had a DEXA scan

* Has had a DEXA scan

Exclusion Criteria:

* Unable to complete DEXA scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2034-08-01 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess the newest version of TBS software on fracture prediction | 10 years

IPD SHARING:
Plan to Share IPD: Undecided